CLINICAL TRIAL: NCT05903885
Title: Using a Cross-sectional Partnership to Improve Prevention and Health Equity Among African Americans
Brief Title: A Cross-sectional Partnership to Improve Prevention and Health Equity Among African Americans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0115-23-EP
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer; Prevention
Keywords: Prevention; Department of motor vehicles; Cross-sectoral partnership; African Americans; Screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The study aims to enroll 600 participants to each of two groups to evaluate strategies in improving colorectal cancer screening rates among African Americans. The groups are the on-site group and the on-site group with social media advertising. The latter group will have exposure to targeted ads on Facebook, Instagram, and YouTube which will run from August 19 to October 29, 2024. The social media campaign will target African American residents of Omaha, aged 45-75. Both groups will be given fecal immunochemical test (FIT) kits, a prepaid return envelope, and an educational brochure when visiting the Department of Motor Vehicles (DMV), 4606 N 56th St Suite 100, Omaha, NE 68104. Both groups will also be given reminder messages and post-FIT navigation support, if needed. Participants' information and perceptions will be collected via surveys. FIT return rate, positive screening rate, and follow-up colonoscopy completion rate will be compared between groups, controlling for covariates.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- On-site Group (Experimental): The on-site distribution group will receive the Fecal Immunochemical Test (FIT) kits directly while visiting the Department of Motor Vehicles (DMV) location at 4606 N 56th St Suite 100, Omaha, NE 68104.
  Participants in the on-site group will be guided through the kit process by trained research staff present. They will be given instructions on collecting the stool sample and using the FIT kit properly.
  They will also be given a culturally tailored educational brochure, a prepaid return envelope, and receive reminder text messages and phone calls within 3 weeks of receipt of the FIT kit. Post-FIT navigation support will be provided for those with positive results or without a family doctor/insurance.
  Interventions: Other: On-site Fecal Immunochemical Test (FIT) Kit Distribution
- On-site Group With Social Media Advertising (Active Comparator): The onsite group with social media advertising participants will receive FIT kits directly at the Department of Motor Vehicles (DMV) location at 4606 N 56th St Suite 100, Omaha, NE 68104. Additionally, they will be exposed to targeted social media advertisements on Facebook, Instagram, and YouTube.
  These participants will encounter ads featuring video content with community member testimonials, emphasizing the importance of colorectal cancer screening for African Americans aged 45-75. The campaign will run from August 19 to October 29, 2024.
  Participants in this group will receive the FIT kits at the DMV along with detailed instructions on how to collect the stool sample and use the kit. They will also receive a culturally tailored educational brochure, prepaid return envelope, reminder text messages, and phone calls within three weeks of receipt of the FIT kit. Post-FIT navigation support will be provided for those with positive results or without a family doctor/insurance.
  Interventions: Other: On-site With Social Media Advertising Fecal Immunochemical Test (FIT) Kit Distribution

INTERVENTIONS:
Other: On-site Fecal Immunochemical Test (FIT) Kit Distribution — Participants will receive home based Fecal Immunochemical Test (FIT) kit directly at the Department of Motor Vehicles (DMV) location at 4606 N 56th St Suite 100, Omaha, NE 68104, by research staff.
  Other Names: Face-to-face distribution
  Arms: On-site Group
Other: On-site With Social Media Advertising Fecal Immunochemical Test (FIT) Kit Distribution — Participants will receive home-based Fecal Immunochemical Test (FIT) kits directly at the Department of Motor Vehicles (DMV) location at 4606 N 56th St Suite 100, Omaha, NE 68104, by research staff supplemented by exposure to targeted social media advertisements.
  Arms: On-site Group With Social Media Advertising

SUMMARY:
African Americans face racial disparities in colorectal cancer (CRC), with lower screening rates and higher incidence and mortality rates. To address this gap and improve CRC screening rates, investigators aims to recruit a total of 1,200 African American participants aged 45-75 during their visits to the DMV, 4606 N 56th St Ste100, Omaha, for CRC screening. All participants will receive a free Fecal Immunochemical Test (FIT) kit with a prepaid return envelope, a culturally tailored educational brochure, reminder text messages and calls, and post-FIT navigation support for participants with positive results or without family doctor/insurance. Kits are returned to a designated Nebraska Medicine lab for testing, and test results will be mailed to participants within 14-21 days. Participants will be assigned to one of two groups: the on-site distribution group or the on-site distribution group with social media advertising group. The social media advertising group will additionally be exposed to targeted ads on platforms like Facebook, Instagram, and YouTube to increase awareness and potentially improve participation rates. The study will compare FIT kit return rates, positive screening rates, and completion rates of follow-up colonoscopies after positive FIT results between the two groups.

DETAILED DESCRIPTION:
African Americans face racial disparities in colorectal cancer (CRC), with lower screening rates and higher incidence and mortality rates. The American Cancer Society reported that African Americans are about 20% more likely to have CRC and 40% more likely to die from it compared to other racial groups. The main reasons for high CRC incidence and mortality for African Americans are structural barriers in access to quality healthcare and timely screening that can be attributed in large part to historical and persistent structural racism in the U.S. To address this gap and improve CRC screening rates among African Americans, this study will partner with the Department of Motor Vehicles (DMV) to recruit African Americans eligible for CRC screening during their regular visits to the DMV. Investigators will recruit 1,200 participants aged 45-75 for CRC screening.

Upon consent, participants' demographic and screening-related information will be collected via a paper-based registration survey (e.g., name, age, gender, race/ethnicity, address, healthcare access, recent CRC screening history, smoking status, and personal/family history of CRC). All participants will receive a free Fecal Immunochemical Test (FIT) kit with a prepaid return envelope, a culturally tailored educational brochure, reminder text messages and calls. Participants will be assigned to one of two groups: the on-site distribution group or the on-site distribution group with social media advertising group. The social media advertising group will additionally be exposed to targeted ads on platforms like Facebook, Instagram, and YouTube from August 19, 2024, to October 29, 2024, to increase awareness and potentially improve participation rates.

Kits are returned to a designated Nebraska Medicine lab, and test results will be mailed to participants within 14-21 days. Follow-up services, including assistance with scheduling colonoscopies and applying for financial support programs, will be provided by a health navigator at Charles Drew Health Center for participants with positive results or those without health insurance or a primary care provider. Outcomes (screening completion rate and positive results) will be compared between the onsite and onsite with social media advertising groups, controlling for other covariates (age, gender, income, previous screening, smoking status, healthcare access, and health beliefs). The study will also assess the cost-effectiveness of each strategy and the completion rate of follow-up colonoscopies after receiving positive FIT results. Participants' perceptions and beliefs about screening will be collected via an online survey.

ELIGIBILITY:
Inclusion Criteria:

* Self-identification as Black or African American
* Between 45 and 75 years old
* Not up-to-date with colorectal cancer (CRC) screening per guidelines
* Willingness to provide contact information for follow-up
* Ability to speak, read, and write English
* Current residency in Douglas County, NE.

Exclusion Criteria:

* History of colorectal cancer (CRC)
* History of adenomas (precancerous polyps) or inflammatory bowel disease
* Family history of colorectal cancer (CRC)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Fecal Immunochemical Test Kit Return Rate | 6 months from date of FIT distribution
  The fecal immunochemical test kit (FIT) return rate is the proportion of participants who have completed the screening by returning the FIT kits.

SECONDARY OUTCOMES:
Fecal Immunochemical Test (FIT) Kit Positive Rate | 6 months from date of FIT distribution
  The fecal immunochemical test (FIT) kit positive rate is the proportion of participants who have positive FIT kit results.
Follow-up Colonoscopy Completion Rate | 6 months from date of positive FIT result notification
  The follow-up colonoscopy completion rate is the proportion of participants with positive FIT results who complete a follow-up colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Jungyoon Kim, PhD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - Department of Motor Vehicles (DMV), Omaha, Nebraska
  - Douglas County Treasurer's Office, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Viale PH. The American Cancer Society's Facts & Figures: 2020 Edition. J Adv Pract Oncol. 2020 Mar;11(2):135-136. doi: 10.6004/jadpro.2020.11.2.1. Epub 2020 Mar 1. No abstract available. PMID 33532112
- [Background] American Cancer Society. Colorectal Cancer Facts and Figures 2020-2022. Atlanta, GA: 2022.
- [Background] American Cancer Society. Key Statistics for Colorectal Cancer. 2022 [updated 1/12/2022; cited 2022 5/2]; Available from: https://www.cancer.org/cancer/colon-rectal-cancer/about/key-statistics.html
- [Background] Mariotto AB, Yabroff KR, Shao Y, Feuer EJ, Brown ML. Projections of the cost of cancer care in the United States: 2010-2020. J Natl Cancer Inst. 2011 Jan 19;103(2):117-28. doi: 10.1093/jnci/djq495. Epub 2011 Jan 12. PMID 21228314
- [Background] Chen CT, Li L, Brooks G, Hassett M, Schrag D. Medicare Spending for Breast, Prostate, Lung, and Colorectal Cancer Patients in the Year of Diagnosis and Year of Death. Health Serv Res. 2018 Aug;53(4):2118-2132. doi: 10.1111/1475-6773.12745. Epub 2017 Jul 26. PMID 28748564
- [Background] Whitlock EP, Lin JS, Liles E, Beil TL, Fu R. Screening for colorectal cancer: a targeted, updated systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2008 Nov 4;149(9):638-58. doi: 10.7326/0003-4819-149-9-200811040-00245. Epub 2008 Oct 6. PMID 18838718
- [Background] US Preventive Services Task Force; Bibbins-Domingo K, Grossman DC, Curry SJ, Davidson KW, Epling JW Jr, Garcia FAR, Gillman MW, Harper DM, Kemper AR, Krist AH, Kurth AE, Landefeld CS, Mangione CM, Owens DK, Phillips WR, Phipps MG, Pignone MP, Siu AL. Screening for Colorectal Cancer: US Preventive Services Task Force Recommendation Statement. JAMA. 2016 Jun 21;315(23):2564-2575. doi: 10.1001/jama.2016.5989. PMID 27304597
- [Background] Wender RC, Doroshenk M, Brooks D, Hotz J, Smith RA. Creating and Implementing a National Public Health Campaign: The American Cancer Society's and National Colorectal Cancer Roundtable's 80% by 2018 Initiative. Am J Gastroenterol. 2018 Dec;113(12):1739-1741. doi: 10.1038/s41395-018-0384-1. Epub 2018 Nov 9. No abstract available. PMID 30413821
- [Background] National Cancer Institute. State Cancer Profiles: 2022.
- [Background] Issaka RB, Taylor P, Baxi A, Inadomi JM, Ramsey SD, Roth J. Model-Based Estimation of Colorectal Cancer Screening and Outcomes During the COVID-19 Pandemic. JAMA Netw Open. 2021 Apr 1;4(4):e216454. doi: 10.1001/jamanetworkopen.2021.6454. PMID 33843997
- [Background] American Cancer Society. Colorectal Cancer Rates Higher in African Americans, Rising in Younger People. 2020 [cited 2022 5/2]; Available from https://www.cancer.org/latest-news/colorectal-cancer-rates-higher-in-african-americans-rising-in-younger-people.html#:~:text=Colorectal%20cancer%20also%20disproportionately%20affects,it%20than%20most%20other%20groups
- [Background] Fedewa SA, Flanders WD, Ward KC, Lin CC, Jemal A, Goding Sauer A, Doubeni CA, Goodman M. Racial and Ethnic Disparities in Interval Colorectal Cancer Incidence: A Population-Based Cohort Study. Ann Intern Med. 2017 Jun 20;166(12):857-866. doi: 10.7326/M16-1154. Epub 2017 May 23. PMID 28531909
- [Background] Laiyemo AO, Doubeni C, Pinsky PF, Doria-Rose VP, Bresalier R, Lamerato LE, Crawford ED, Kvale P, Fouad M, Hickey T, Riley T, Weissfeld J, Schoen RE, Marcus PM, Prorok PC, Berg CD. Race and colorectal cancer disparities: health-care utilization vs different cancer susceptibilities. J Natl Cancer Inst. 2010 Apr 21;102(8):538-46. doi: 10.1093/jnci/djq068. Epub 2010 Mar 31. PMID 20357245
- [Background] Office of the Assistant Secretary for Planning and Evaluation, U.S. Department of Health and Human Services. Health Insurance Coverage and Access to Care Among Black Americans: Recent Trends and Key Challenges. (Issue Brief No. HP-2022-07). February 2022.
- [Background] White A, Thompson TD, White MC, Sabatino SA, de Moor J, Doria-Rose PV, Geiger AM, Richardson LC. Cancer Screening Test Use - United States, 2015. MMWR Morb Mortal Wkly Rep. 2017 Mar 3;66(8):201-206. doi: 10.15585/mmwr.mm6608a1. PMID 28253225
- [Background] Horne HN, Phelan-Emrick DF, Pollack CE, Markakis D, Wenzel J, Ahmed S, Garza MA, Shapiro GR, Bone LR, Johnson LB, Ford JG. Effect of patient navigation on colorectal cancer screening in a community-based randomized controlled trial of urban African American adults. Cancer Causes Control. 2015 Feb;26(2):239-246. doi: 10.1007/s10552-014-0505-0. Epub 2014 Dec 17. PMID 25516073
- [Background] Christy SM, Davis SN, Williams KR, Zhao X, Govindaraju SK, Quinn GP, Vadaparampil ST, Lin HY, Sutton SK, Roethzeim RR, Shibata D, Meade CD, Gwede CK. A community-based trial of educational interventions with fecal immunochemical tests for colorectal cancer screening uptake among blacks in community settings. Cancer. 2016 Nov 15;122(21):3288-3296. doi: 10.1002/cncr.30207. Epub 2016 Jul 15. PMID 27420119
- [Background] Campbell MK, James A, Hudson MA, Carr C, Jackson E, Oakes V, Demissie S, Farrell D, Tessaro I. Improving multiple behaviors for colorectal cancer prevention among african american church members. Health Psychol. 2004 Sep;23(5):492-502. doi: 10.1037/0278-6133.23.5.492. PMID 15367069
- [Background] Holt CL, Litaker MS, Scarinci IC, Debnam KJ, McDavid C, McNeal SF, Eloubeidi MA, Crowther M, Bolland J, Martin MY. Spiritually based intervention to increase colorectal cancer screening among African Americans: screening and theory-based outcomes from a randomized trial. Health Educ Behav. 2013 Aug;40(4):458-68. doi: 10.1177/1090198112459651. Epub 2012 Oct 2. PMID 23033548
- [Background] Powe BD, Ntekop E, Barron M. An intervention study to increase colorectal cancer knowledge and screening among community elders. Public Health Nurs. 2004 Sep-Oct;21(5):435-42. doi: 10.1111/j.0737-1209.2004.21507.x. PMID 15363024
- [Background] Nebraska Department of Motor Vehicles. 2021 Annual Report. 2021.
- [Background] Harrison TR, Morgan SE, Di Corcia MJ. Effects of information, education, and communication training about organ donation for gatekeepers: clerks at the Department of Motor Vehicles and organ donor registries. Prog Transplant. 2008 Dec;18(4):301-9. doi: 10.1177/152692480801800414. PMID 19186584
- [Background] Denberg TD, Melhado TV, Coombes JM, Beaty BL, Berman K, Byers TE, Marcus AC, Steiner JF, Ahnen DJ. Predictors of nonadherence to screening colonoscopy. J Gen Intern Med. 2005 Nov;20(11):989-95. doi: 10.1111/j.1525-1497.2005.00164.x. PMID 16307622
- [Background] Bailey JR, Aggarwal A, Imperiale TF. Colorectal Cancer Screening: Stool DNA and Other Noninvasive Modalities. Gut Liver. 2016 Mar;10(2):204-11. doi: 10.5009/gnl15420. PMID 26934885
- [Background] Goodwin BC, Ireland MJ, March S, Myers L, Crawford-Williams F, Chambers SK, Aitken JF, Dunn J. Strategies for increasing participation in mail-out colorectal cancer screening programs: a systematic review and meta-analysis. Syst Rev. 2019 Nov 4;8(1):257. doi: 10.1186/s13643-019-1170-x. PMID 31685010
- [Background] Davis MM, Freeman M, Shannon J, Coronado GD, Stange KC, Guise JM, Wheeler SB, Buckley DI. A systematic review of clinic and community intervention to increase fecal testing for colorectal cancer in rural and low-income populations in the United States - How, what and when? BMC Cancer. 2018 Jan 6;18(1):40. doi: 10.1186/s12885-017-3813-4. PMID 29304835
- [Background] Jager M, Demb J, Asghar A, Selby K, Mello EM, Heskett KM, Lieberman AJ, Geng Z, Bharti B, Singh S, Gupta S. Mailed Outreach Is Superior to Usual Care Alone for Colorectal Cancer Screening in the USA: A Systematic Review and Meta-analysis. Dig Dis Sci. 2019 Sep;64(9):2489-2496. doi: 10.1007/s10620-019-05587-6. Epub 2019 Mar 26. PMID 30915656
- [Background] Jean-Jacques M, Kaleba EO, Gatta JL, Gracia G, Ryan ER, Choucair BN. Program to improve colorectal cancer screening in a low-income, racially diverse population: a randomized controlled trial. Ann Fam Med. 2012 Sep-Oct;10(5):412-7. doi: 10.1370/afm.1381. PMID 22966104
- [Background] Roy S, Dickey S, Wang HL, Washington A, Polo R, Gwede CK, Luque JS. Systematic Review of Interventions to Increase Stool Blood Colorectal Cancer Screening in African Americans. J Community Health. 2021 Feb;46(1):232-244. doi: 10.1007/s10900-020-00867-z. PMID 32583358